CLINICAL TRIAL: NCT04565288
Title: Enhancing the Effects of Adolescent Alcohol Treatment With Atomoxetine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1805002051; K24AA026326 (NIH)
Record Dates: First submitted 2020-08-28; First posted 2020-09-25 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atomoxetine (Experimental): Atomoxetine (40 mg/day for 3 days then 80 mg/day thereafter) during a 6-week medication trial
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Identical matching placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Participants randomized to receive the study medication, atomoxetine (brand name: Straterra) for 6-weeks (40 mg/day for 3 days then 80 mg/day thereafter). A comparator group will receive placebo (sugar pills).
  Other Names: Strattera
  Arms: Atomoxetine
Drug: Placebo — Matching placebo (sugar pill)
  Arms: Placebo

SUMMARY:
The primary objectives of this study are twofold. The first primary objective is to evaluate the feasibility, acceptability, and tolerability of atomoxetine (40 mg/day for 3 days then 80 mg/day thereafter) as compared to placebo for 6 weeks plus a psychosocial platform comprised of motivational enhancement therapy and cognitive behavioral therapy (MET-CBT) among adolescents (ages 14 to 19 years) with alcohol use disorder as confirmed by the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5™). The second primary objective is to leverage a human laboratory paradigm and ecological momentary assessment (EMA) methods to evaluate the effects of atomoxetine on intermediate phenotypes associated with alcohol use and outcomes in clinical trials.

DETAILED DESCRIPTION:
This proof-of-concept study is a double-blind, randomized, placebo-controlled, parallel-group, single-site study designed to assess the feasibility, acceptability, and tolerability of atomoxetine for alcohol use disorder among adolescents ages 14 to 19 years. In addition, this project will test the effects of atomoxetine, as compared with placebo, on responses to in vivo alcohol cue exposure in the human laboratory setting. After obtaining consent/parent permission/assent, youth and, if younger than 18 years, their parent will complete a medical history interview to screen for eligibility. Youth will also be screened for eligibility. If eligible for the study, participants will be randomized in an approximate 1:1 ratio (targeting 21 participants per group - 42 participants total) to either atomoxetine or placebo for 6 weeks. Atomoxetine will be dosed at 40 mg/day for three days then increased to the maintenance dose of 80 mg (active) taken orally once daily (QD) for an additional 5.5 weeks. Participants randomized to the placebo condition will be given an equal number of visually matched capsules.

Participants will be seen in the clinic at the in-person screening appointment, the randomization/baseline session, and at 8 other times during the study. Three follow-up telephone interviews will occur at 2 weeks and three and six months after the last in-clinic visit. At the randomization/baseline visit and after 4 weeks of investigational product administration (i.e., Study Week 7), participants will undergo a human laboratory paradigm (i.e., alcohol cue reactivity assessment). In addition, participants will complete EMA on a smartphone throughout the day in their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14 to 20 years, inclusive
* Self-reports consuming alcohol ≥ 2 days/week on average in the past 28 days
* Meets the DSM-5 criteria for alcohol use disorder (AUD)
* Interested in reducing alcohol use
* Be able to verbalize an understanding of the consent/assent form, able to provide written informed consent/assent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English, and able to complete the questionnaires required by the protocol.
* If younger than 18 years, parent permissions is required.
* Be able to take oral medication and be willing to adhere to the medication regimen
* Complete all assessments required at screening and baseline
* Provide contact information of someone, such as a parent or other family member, who may be able to contact the subject in case of a missed clinic appointment or follow-up assessment.
* Be someone who in the opinion of the investigator would be expected to complete the study protocol
* Agree to the schedule of visits, verbally acknowledge that s/he will be able to attend each scheduled visit, participate in phone visits and that s/he does not have any already scheduled events or a job that may substantially interfere with study participation.
* Not anticipate any significant problems with transportation arrangements or available time to travel to the study site over the next 2 months.
* Agree (if the subject is female and of child bearing potential) to use birth control

Exclusion Criteria:

* Currently receiving treatment for AUD
* Significant alcohol withdrawal symptoms
* Coexisting moderate to severe substance use disorder other than cannabis and nicotine
* Urine toxicology screen positive drugs of abuse except for cannabis
* Treated with pharmacotherapy for AUD or a carbonic anhydrase inhibitor in past 30 days
* Compelled to alcohol treatment by the juvenile justice system or has probation or parole requirements that might interfere with study participation
* History of liver disease or have clinically significant abnormal laboratory values
* History of renal impairment or renal stones, narrow angle glaucoma or pheochromocytoma, heart problems or defects, abnormal blood pressure, progressive neurodegenerative disorder, or clinically significant neurological disorders
* Clinically significant physical abnormalities per physical exam, hematological assessment, bilirubin concentration, or urinalysis
* Pregnancy, nursing, or refusal to use reliable birth control, if female
* Psychotropic medication use in the past 30 days
* Current or lifetime diagnosis of psychotic disorders
* Current bipolar disorder
* Current major depressive episode
* Ever attempted suicide
* Current (past year) suicidality risk
* Known sensitivity to atomoxetine
* Be anyone who in the opinion of the investigator could not be safely withdrawn from alcohol without medical detoxification
* Serious or unstable medical illness or any potentially life-threatening or progressive medical condition other than addiction that may compromise subject safety or study conduct
* Abnormal calculated creatinine clearance defined as < 80 mL/min
* Evidence of cirrhosis of the liver (albumin < 3.2 g/dL, or ascites by physical exam)

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miranda, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded into the appropriate NIH repository as required.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: Within 12-months of publication
Access Criteria: Any investigator who requests access in writing will be provided with the requested information.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 21 | 21
Completed | 17 | 18
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.8 (0.8) | 18.9 (0.7) | 18.9 (.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 13 | 15 | 28
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Days Abstinent from Alcohol (% of Days) [Mean (Standard Deviation); unit: Percent of Days] — This measure describes the percentage of days participants consumed alcohol during the 28 days before the baseline assessment session. This measure characterizes the sample's alcohol use at baseline, before randomization to atomoxetine or placebo.
  Percent of Days | 65.65 (10.26) | 61.57 (16.67) | 63.61 (13.82)
Number of Standard Alcohol Drinks per Drinking Day [Mean (Standard Deviation); unit: Drinks per Drinking Day] — This measure describes the number of drinks that participants consumed per drinking day during the 28 days preceding the baseline assessment session. This measure characterizes the sample's alcohol use at baseline, before randomization to atomoxetine or placebo.
  Drinks per Drinking Day | 5.57 (2.45) | 4.72 (1.96) | 5.14 (2.23)
Heavy Drinking Days (%) [Mean (Standard Deviation); unit: Percent of Days] — This measure describes the percentage of days participants engaged in heavy drinking, defined as 4 or more drinks per day for females and 5 or more drinks per day for males, during the 28 days before the baseline assessment session. This measure characterizes the sample's alcohol use at baseline, before randomization to atomoxetine or placebo.
  Percent of Days | 26.02 (10.69) | 27.89 (12.61) | 26.96 (12.05)

OUTCOME MEASURES:

1. Primary Outcome: Completion Rates
Description: Number and percentage of youth who complete the active medication phase will determine feasibility.
Time Frame: 6-week active treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 21 | 21
Participants | 17 | 18

2. Primary Outcome: Number of Participants Who Rate Their Treatment Experience in the "Satisfactory" or "Highly Satisfactory" Range on the CSQ-8
Description: The Client Satisfaction Questionnaire (CSQ-8), which ranges in scores from 8 to 32 (higher scores indicate higher satisfaction), will determine acceptability. Treatment satisfaction will be considered acceptable if the number and percentage of subjects who rate their treatment experience in the "satisfactory" or "highly satisfactory" range on the CSQ-8 is ≥ 80%.
Time Frame: 6-week active treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 21 | 21
Participants | 21 | 19

3. Secondary Outcome: Alcohol Craving
Description: The primary measure of alcohol craving is the number and percentage of participants who report any level of alcohol craving during a laboratory alcohol-cue exposure paradigm using the following single item: How strong is your craving to drink alcohol? Scores range from 0 (None) to 20 (Extremely Strong). Individuals who endorse any level of alcohol craving (e.g., > 1) are considered to experience craving. Individuals who do not report any alcohol craving (e.g., 0) will be regarded as non-craving.
Time Frame: Alcohol craving was assessed during a laboratory alcohol-cue exposure paradigm, at week 5. Participants rated their alcohol craving immediately following exposure to alcohol and water cues. The outcomes measure is craving after alcohol cue exposure.
Measure: Count of Participants; unit: Participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 11 | 18
Participants | 5 | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 6-week treatment period.
Description: Adverse events were captured using criteria set forth by the U.S. Food and Drug Adminisration (FDA)
Arm/Group | Atomoxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 19/21 | 19/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=21) | Placebo (N=21)
Nausea (Gastrointestinal disorders) | 9 | 8
Hypertension (Cardiac disorders) | 8 | 6
Headache (General disorders) | 7 | 7
Flu-like symptoms (General disorders) | 4 | 5
Insomnia (General disorders) | 4 | 3
Sore throat (General disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Nasal congestion (General disorders) | 1 | 4
Decreased appetite (Gastrointestinal disorders) | 2 | 2
Drowsiness (General disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 3 | 0
Fever (General disorders) | 2 | 1
Stomach pain (Gastrointestinal disorders) | 2 | 1
Tingling (General disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0
Weight gain (Metabolism and nutrition disorders) | 0 | 3
Heart racing (Cardiac disorders) | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The purpose of this preliminary pilot trial was to establish the feasibility and acceptability of atomoxetine for treating alcohol use disorder among adolescents. The findings do not address whether this medication is efficacious for this purpose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT04565288/Prot_SAP_002.pdf
  • Informed Consent Form (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT04565288/ICF_001.pdf